CLINICAL TRIAL: NCT03559153
Title: Effect of Passive and Active Rest Break in Musculoskeletal Complains in Office Workers
Brief Title: Effect of Passive and Active Rest Break in Musculoskeletal Complains
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Cidade de Sao Paulo (Other)
Responsible Party: Principal Investigator, Rosimeire Simprini Padula, PhD. Clinical Professor, Universidade Cidade de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1.736.249
Record Dates: First submitted 2018-04-29; First posted 2018-06-15 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Occupational Diseases; Work-related Injury
Keywords: Office workers; Worker health; Work ability; Musculoskeletal disease
MeSH Terms: conditions — Occupational Diseases; Musculoskeletal Diseases | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): All workers will receive ergonomics instructions. Instruction for rest break.
- Passive rest break - Shiatsu massage (Experimental): All workers will receive ergonomics instructions. The workers will be receive "quick massage" using shiatsu techniques.
  Interventions: Other: Shiatsu massage
- Active rest break - Physical Exercise Program (Active Comparator): All workers will receive ergonomics instructions. The workers will be receive exercises during the rest break.
  Interventions: Other: Physical Exercise

INTERVENTIONS:
Other: Shiatsu massage — The shiatsu massage will be during the rest break by 15 minutes.
  Arms: Passive rest break - Shiatsu massage
Other: Physical Exercise — The Physical Exercise will be during the rest break by 15 minutes.
  Arms: Active rest break - Physical Exercise Program

SUMMARY:
Work-related musculoskeletal disorders are highly disabling. Therefore, finding preventive solutions is fundamental, in order to reduce the damages to workers and society. Therefore the objective of this study will be to evaluate the effect of passive and active pauses in the control of musculoskeletal complaints of office workers. This is a randomized controlled trial by cluster, which will be performed with 286 office workers (administrative sectors). Employees with physical disabilities will not be included in the study. The workers will be distributed into three groups: active control group, and the two intervention groups massage and workout gymnastics. The active control group and the other groups will be guidelines on ergonomic adjustments of the work station, and performing a 10-minute break every 50 minutes work. The intervention groups (passive and active) will receive different interventions: group massage in the chair and group gymnastics labor. The massage will be performed 2x per week for 10 minutes, and workout 2x per week for 15-20minutes. The primary outcomes assessed will be musculoskeletal complaints of pain intensity. And as a secondary outcome will be the ability to work, perception of ergonomic risk factors, psychosocial factors and fatigue, level of physical activity. Outcomes will be assessed at baseline and after 4 months. It is expected that exercise intervention (active pause) is more effective than passive pause (massage), and that pause and guidance can reduce musculoskeletal complaints, pain intensity, and other outcomes evaluated.

DETAILED DESCRIPTION:
Inclusion and Exclusion Criteria Office workers, who work at least 6 hours a day in a sitting position, will be included. disabled employees will not be included.

Sample size: The prevalence of complaints and pain intensity in the arm, neck and shoulder regions, in addition to the lumbar region. A statistical power of 80%, α = 5%, sample loss of 15% will be considered for the sample calculation. The reduction expected of the prevalence of musculoskeletal complaints and pain will be 20%. Therefore, it will be necessary to perform the study 286 workers, allocated in control group (CG), intervention groups (IG), passive rest break - Shiatsu - Quick massage (SGM); and comparative group using active rest break - Compensatory exercise program(CE).

the outcomes will be evaluated at the individual level, since they reflect aspects of workers' health. Data on outcome measures will be assessed at baseline and after 4 months. After a period of 4 months, the sector that received only a break or massage can receive work gymnastics, if the hypothesis of this study is confirmed on the effectiveness of the exercise on the other interventions. Both groups of workers will be followed up in a longitudinal study in subsequent months and compared to the other workers identified, within the established criteria for risk analysis, for 4 months.

Primary outcome: The occurrence of musculoskeletal symptoms (pain, tingling or numbness) will be evaluated by means of the Nordic Questionnaire for Musculoskeletal Symptoms The intensity of the pain will be evaluated by the Verbal Numerical Scale of Pain23. It is an 11-point scale, in which 0 means "no pain" and 10 means "worst possible pain".

Secondary outcomes: 1) Work ability index (WAI) to identify the worker's perception at the moment or in the near future; 2)

ELIGIBILITY:
Inclusion Criteria:

* Office workers, who work at least six hours a day in a sitting position, will be included.

Exclusion Criteria:

* Physical disability employees will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2019-01-20 (Actual); Study Completion 2019-03-03 (Actual)

PRIMARY OUTCOMES:
Change from Musculoskeletal complains at 4,8,12,16 weeks | At baseline, and after 4, 8, 12, and 16 weeks
  The occurrence of musculoskeletal symptoms (pain, tingling or numbness) will be evaluated through the Nordic Questionnaire for Musculoskeletal Symptoms (QNSO). The interviewee will answer simple questions (yes or no) regarding the musculoskeletal symptoms he has experienced in the last 12 months and / or the last 7 days, the occurrence of functional incapacity and the demand for help from a health professional in the last 12 months resulting from these symptoms.
Change from Pain Intensity at 4, 8, 12, 16 weeks | At baseline and after 4, 8, 12, and 16 weeks
  The intensity of the pain will be evaluated by the Verbal Numerical Scale of Pain. It is an 11-point scale, in which 0 means "no pain" and 10 means "worst possible pain".

SECONDARY OUTCOMES:
Change from Work Ability Index (WAI) at 16 weeks | At baseline and after 16 weeks
  The Work Ability Index (WAI) is an instrument that evaluates the worker's perception of how well he or she is or will be at the moment or in the near future and how well he can perform his or her job, depending on the requirements, of their state of health and physical and mental capacities.

CONTACTS AND LOCATIONS:
Locations (1):
- Rosimeire Simprini Padula, Atibaia, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided